CLINICAL TRIAL: NCT05054387
Title: A Phase 4, Open Label, Safety and Efficacy Study of Fabrazyme® (Agalsidase Beta) as Enzyme Replacement Therapy in Chinese Participants With Fabry Disease
Brief Title: China Post-marketing Surveillance (PMS) Study of Fabrazyme®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS16583; U1111-1255-4881 (Registry Identifier: UTN)
Record Dates: First submitted 2021-09-09; First posted 2021-09-23 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Agalsidase beta (Experimental): Agalsidase beta treatment at approved dose and regimen, administered once every 2 weeks as an IV infusion
  Interventions: Drug: Agalsidase beta

INTERVENTIONS:
Drug: Agalsidase beta — Powder for concentration into a solution Intravenous (IV) infusion
  Other Names: GZ419828 Fabrazyme

SUMMARY:
This is a 54-week Phase 4, open label, single arm study to evaluate the safety and the efficacy of Fabrazyme (agalsidase beta) as enzyme replacement therapy (ERT) in Chinese participants with Fabry Disease.

DETAILED DESCRIPTION:
Study participation for each patient will be total of 54 weeks which will include 4 weeks of screening, 48 weeks of treatment period and 2 weeks of post study treatment observation

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 8 years of age or older, at the time of signing the informed consent
* Participants naive to agalsidase beta and agalsidase alpha
* Chinese participants diagnosed with Fabry disease and with documented plasma or leukocyte αGAL activity deficient below laboratory's reference range, and/or documented diagnosis by genotyping
* Participants must have one or more symptoms and signs consistent with manifestations of Fabry disease (not limited to neuropathic pain, chronic kidney disease, hypertrophic cardiomyopathy, cardiac rhythm disturbances, cerebrovascular involvement, cornea verticillata, angiokeratoma, gastrointestinal symptoms, hypo- or anhydrosis)
* A female participant is eligible to participate if she is not pregnant or breastfeeding and use an acceptable contraceptive method
* Participants and/or participant's legal representative capable of giving signed informed consent.

Exclusion Criteria:

* The participant has undergone kidney transplantation.
* The participant has a clinically significant organic disease (with the exception of symptoms relating to Fabry disease) in the opinion of the Investigator, would preclude participation in the trial.
* Received an investigational drug, or device, other than Fabrazyme, within 30 days of anticipated IMPs administration or 5 half-lives of the previous investigational drug, whichever is longer.
* The patient has current evidence of kidney failure or renal insufficiency, as defined by eGFR <30 mL/min/1.73 m2.
* Individuals who have life threatening hypersensitivity (anaphylactic reaction) to the active substance or any of the excipients included.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) | Baseline to week 50
  Including TEAE, SAEs, and adverse events of special interest (AESIs) including infusion associated reactions (IARs) and change of clinical laboratory, vital signs and ECG

SECONDARY OUTCOMES:
The absolute changes of plasma globotriaosylsphingosine (lyso-GL3) | from baseline to Week 6, Week 12, Week 24 and Week 48
The percent changes of plasma lyso-GL3 | from baseline to Week 6, Week 12, Week 24 and Week 48
The absolute changes of plasma globotriaosylceramide (GL3) | from baseline to Week 6, Week 12, Week 24 and Week 48
The percent changes of plasma GL3 | from baseline to Week 6, Week 12, Week 24 and Week 48
The number of participants with abnormal plasma GL3 values per central lab reference range | at Week 6, Week 12, Week 24 and Week 48
The percentage of participants with abnormal plasma GL3 values per central lab reference range | at Week 6, Week 12, Week 24 and Week 48
The change of Fabry disease symptoms | from baseline to Week 24 and Week 48
  The change of Fabry disease symptoms assessment (improved, worsen or same): angiokeratoma, sweating, chronic abdominal pain, level of activity, exercise tolerance and heat tolerance, headache, tinnitus
The absolute change of estimated glomerular filtration rate (eGFR) by chronic kidney disease epidemiology collaboration (CKD-EPI) for adult (≥18 years) | from baseline to Week 12, Week 24, Week 36 and Week 48
The absolute change of estimated glomerular filtration rate (eGFR) by Schwartz for children (8 ≤age <18 years) | from baseline to Week 12, Week 24, Week 36 and Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- China (6):
  - Investigational Site Number :1560003, Beijing
  - Investigational Site Number :1560002, Beijing
  - Investigational Site Number :1560001, Shanghai
  - Investigational Site Number :1560004, Shanghai
  - Investigational Site Number :1560006, Taiyuan
  - Investigational Site Number :1560005, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Ren H, Zhang W, Ouyang Y, Guo J, Xu H, Ma J, Luo X, Pan X, Yuan Y, Zhang W, Shen Q, Li B, Feng Q, Liu S, Chen N. A phase 4, open-label, multicenter study of the safety and efficacy of agalsidase beta in Chinese patients with Fabry disease. Orphanet J Rare Dis. 2025 Aug 4;20(1):401. doi: 10.1186/s13023-025-03950-7. PMID 40760696
- See also: LPS16583 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25283&tenant=MT_SNY_9011